CLINICAL TRIAL: NCT04826510
Title: Objective to Evaluate the Efficacy and Safety of Peropirone Hydrochloride Tablets in the Treatment of Adolescent Bipolar Depressive Episode: a Multicenter Open Randomized Controlled Clinical Trial
Brief Title: Efficacy and Safety of Peropirone Hydrochloride Tablets in the Treatment of Adolescent Bipolar Disorder Depression
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3.0
Record Dates: First submitted 2021-01-31; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2020-09

CONDITIONS: Depressive Disorder
MeSH Terms: conditions — Depressive Disorder | interventions — Lithium Carbonate

STUDY DESIGN:
Intervention Model Description: The study is expected in the nine and clinical study of cooperative unit to carry out clinical research network, each is expected to include subjects about 21 cases (7 cases of lithium carbonate group, pp horse of the 7 cases, hydrochloric acid hydrochloric acid lithium carbonate + pp ROM horse lung group of 7 cases), with 189 recruit subjects (lithium carbonate group 63 examples, hydrochloric acid pp ROM horse lung group 63 examples, lithium carbonate + pp hydrochloride horse lung group 63 examples. The study is expected to be completed within two years.
Who Masked: Participant, Outcomes Assessor
Masking Description: Subjects will be randomly assigned to the lithium carbonate group, piperopirone hydrochloride group or the lithium carbonate + Piperopirone hydrochloride group after obtaining the corresponding random number according to the order of inclusion. According to the random centers, the lithium carbonate group: piperopirone hydrochloride group: lithium carbonate + Piperopirone hydrochloride group was 1:1:1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lithium carbonate group (Active Comparator): Lithium carbonate treatment, stable blood lithium concentration 0.5-1.2 mmol / L, course of 8 weeks.
  Interventions: Drug: Lithium Carbonate Pill
- Perospirone hydrochloride group (Experimental): The dosage of perospirone hydrochloride tablets was 16-36 mg / D for 8 weeks.
  Interventions: Drug: Perospirone hydrochloride tablets
- Lithium carbonate + perospirone hydrochloride group (Experimental): The stable blood lithium concentration was 0.5-1.2 mmol / L, and the dose of perospirone hydrochloride tablets was 16-36 mg / D for 8 weeks.
  Interventions: Drug: Lithium carbonate + perospirone hydrochloride

INTERVENTIONS:
Drug: Perospirone hydrochloride tablets — The dosage of perospirone hydrochloride tablets was 16-36 mg / D for 8 weeks.
  Arms: Perospirone hydrochloride group
Drug: Lithium carbonate + perospirone hydrochloride — The stable blood lithium concentration was 0.5-1.2 mmol / L, and the dose of perospirone hydrochloride tablets was 16-36 mg / D for 8 weeks.
  Arms: Lithium carbonate + perospirone hydrochloride group
Drug: Lithium Carbonate Pill — Lithium carbonate treatment, stable blood lithium concentration 0.5-1.2 mmol / L, course of 8 weeks.
  Arms: Lithium carbonate group

SUMMARY:
Bipolar disorder, a type of mood disorder that occurs in various forms, such as depression, mania, hypomania or irregularity.According to the World Health Organization mental health survey, the lifetime prevalence of bipolar disorder is 2.4%; the 12-month prevalence was 1.5%. The lifetime incidence in Shenzhen was 1.5%, and the 12-month incidence was 1.1%. In another study in Hong Kong, the 12-month prevalence of bipolar I, II, and "soft" II was 1.4%, 0.5%, and 1.8%, respectively. Due to endocrine effects, bipolar disorder is more common in women than men, and mainly occurs in late adolescence and early adulthood, with an early trend. An investigation involving 23 countries around the world found that the average age of onset of bipolar disorder was 25 years old, and the low age group (17.24±3.20 years old) accounted for 41.7%. Another study in the United States showed that the average age of onset of bipolar disorder was 20 years old, and the low age group (14.5±4.9 years old) accounted for 63%. With the improvement of medical level, the diagnosis rate of bipolar disorder is getting closer to the true prevalence rate.

Without active treatment, the symptoms of bipolar disorder, especially depression, will accompany the patients for a long time. The quality of life of patients is seriously affected.

The safety of piperopilon hydrochloride has been widely recognized from pre-market clinical research to post-market clinical practice. A total of a clinical study involving 1191 patients showed that the incidence of side effects from long-term use of piperopilone was 21.3%, and the main side effects were mild in the nervous and digestive systems. In addition, it has been reported that piperopirone is also safe and effective for adolescents.Therefore, the investigators designed this study to explore the atypical antipsychotic drug piperopirone as a monotherapy or in combination with mood stabilizer.Clinical efficacy and safety of lithium acid in the treatment of depressive episodes in adolescents with bipolar disorder, and its improvement in cognitive function were assessed.The goal is to evaluate the efficacy and safety of piperopilone hydrochloride tablets in the treatment of bipolar depressive episode in adolescents.

DETAILED DESCRIPTION:
Participants will be randomly assigned to the lithium carbonate group, piperopirone hydrochloride group or the lithium carbonate + Piperopirone hydrochloride group after obtaining the corresponding random number according to the order of inclusion. According to the random centers, the lithium carbonate group: piperopirone hydrochloride group: lithium carbonate + Piperopirone hydrochloride group was 1:1:1

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients or inpatients who met the diagnostic criteria of DSM-5 or ICD-10 for depressive episode of bipolar disorder.
2. Willing to participate in clinical research and sign informed consent
3. 12 ≤ age ≤ 18
4. HAMD-17 score ≥ 17; HAMD-17 item 1 (depression) ≥ 2, and YMRS ≤ 12
5. Physical examination, laboratory examination, vital signs and 12 lead ECG showed that the physical condition was stable. If any test results are beyond the normal range, they can be included only if they are judged to be abnormal or deviated from the normal values but have no clinical significance or belong to reasonable conditions in the study population. Such decisions must be recorded in the subject's original file and signed by the researcher

Exclusion Criteria:

1. Besides bipolar disorder, the diagnosis includes schizophrenia, schizophrenic affective disorder, schizoid disorder, depression, dissociation disorder, borderline personality disorder, material dependence, autism, organic mental disease, etc
2. Other conditions except bipolar disorder were diagnosed, such as schizophrenia, schizophrenic affective disorder, schizophrenia like disorder, depression, dissociation disorder, borderline personality disorder, material dependence, autism, organic mental disease, etc. according to the judgment of the researcher, the patient is at risk of suicide or injury to others, or HAMD-17 item 3 Score ≥ 3, or attempted suicide in the past six months
3. Patients with rapid circulation type;
4. Those who had suffered from serious heart, liver, brain, lung, kidney and other serious diseases in the past or at present, and the researchers considered that they were not suitable for the study;
5. The results of Biochemistry, hematology, electrocardiogram or urine test were not within the normal value range of the laboratory at the time of screening, and had clinical significance according to the judgment of the researchers (except for the abnormal indexes of reasonable condition in the research population, such as abnormal blood glucose and blood lipid indexes);
6. The subjects received electroconvulsive therapy (ECT) within 6 months before enrollment;
7. There was a history of malignant tumor or complications;
8. Known allergy history or complications to test drug or ingredient (with previous history of allergic reaction caused by drug, rash, urticaria, etc.);
9. Pregnant and lactating women and patients unable to take appropriate contraceptive measures during the trial period;
10. Patients with previous suicidal behavior or existing strong suicidal tendency and patients with serious excited and aggressive behavior.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 189 (Estimated)
Dates: Start 2020-11-25 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinical Global Impression Scale-Bipolar Disorder Scale (CGI-BP-S) score | Change from baseline at 2,4,8 week.
  The investigators adopt the clinical General Impression Scale - Bipolar Disorder Scale (CGI-BP-S) score to analyze the scores of the subjects in different periods.
Hamilton Depression Scale (HAMD-17) score | Change from baseline at 2,4,8 week.
  The investigators adopt the Hamilton Depression Scale (HAMD-17) score to judge the subjects' depression. Starting points: Hamilton Depression Scale (HAMD-17)) ≥2, clinical remission: Hamilton Depression Scale (HAMD-17)) <7.

SECONDARY OUTCOMES:
Young's Manic Rating Scale (YMRS) score | Change from baseline at 2,4,8 week.
  Young's Manic Rating Scale (YMRS) was used to determine the degree of mania in the subjects. Initial score: Young's Manic Rating Scale (YMRS) score ≤12; Clinical remission: Young's Manic Rating Scale (YMRS) score ≤5.
Montreal Cognitive Assessment Scale (MoCA) score | Change from baseline at 8 week.
  The investigators adopt the Montreal cognitive assessment scale (MoCA) score to judge whether the subjects with normal cognition and affect its subsequent different drugs.
Wisconsin Card Sorting Test (WCST-128) score | Change from baseline at 8 week.
  The investigators used the Wisconsin Card Sorting Test (WCST-128) score to determine whether the subjects had normal cognition. Reference value: total response number < 60: indicating cognitive abnormalities; Incorrect response number > 45: indicates cognitive abnormality
WISC score for Children | Change from baseline at 8 week.
  WISC Score for Children was used to determine whether subjects' IQ was affected by their disease. Reference value: 1. Low: Total IQ score ≤90; 2. Normal: Total IQ score is 90-110; High IQ: total IQ score ≥110

CONTACTS AND LOCATIONS:
Overall Officials: Yiru Fang, professor, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
After the trial is over, after obtaining the written consent of the sponsor, the research unit can publish the research results of this clinical trial in the form of a paper, but the source of the drug must be stated. The investigator of each research unit has the right to sign the paper. ponsors can also publish papers or use experimental content, or participate in signing
Supporting Information: Study Protocol, CSR
Time Frame: start from 2021.6.30,last for 2years
Access Criteria: the cooperative partners